CLINICAL TRIAL: NCT00152490
Title: A Phase III Multi-national, Multi-centre, Double-blind Placebo-controlled Parallel Group, 26 Week Study to Assess the Safety and Efficacy of the Humanised Anti-TNF PEG Conjugate, CDP870 400 mg sc, (Dosed at Weeks 0, 2, 4 Then 4-weekly to Week 24), in the Treatment of Patients With Active Crohn's Disease
Brief Title: A Study to Test the Effect of CDP870 in the Treatment of Crohn's Disease Over 26 Weeks, Comparing CDP870 to a Dummy Drug (Placebo)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: C87031
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2010-02

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease, CDP870, CDAI, clinical response, remission,; Certolizumab Pegol, Cimzia
MeSH Terms: conditions — Crohn Disease; Anemia, Dyserythropoietic, Congenital | interventions — Certolizumab Pegol

INTERVENTIONS:
Drug: Certolizumab Pegol (CDP870)

SUMMARY:
A 26 week study to examine the efficacy, safety and pharmacokinetics of CDP870 in Crohn's disease

DETAILED DESCRIPTION:
Receiving immunosuppressants (azathioprine/6-MP/methotrexate) at Week 0 or not.

604 patients will be enrolled with 1006 patients screened (to allow for 25% screen failures between screening and Week 0 and expected presentation at Screening of 60% of patients with CRP < 10 mg/L and 40% of patients with CRP ≥ 10 mg/L).

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of Crohn's disease confirmed (at least 3 months prior to study entry) either by radiological, endoscopic or histological evidence, affecting the terminal ileum (L1), colon (L2) or ileocolon (L3*. *Vienna Classification (1998)
* Active Crohn's disease (≥ 220 and ≤ 450) scored over the 7 days prior to the first dose of study drug.
* Male and female aged 18 years or above at screening.
* Patients who meet all concomitant medication criteria in the protocol specified table. For all drugs being taken at screening, the patient should be able to remain on a stable dose throughout the duration of the study, although steroids may be tapered starting at Weeks 8 to 12.

Exclusion Criteria:

* Crohn's Disease Related
* Fistula abscess present at screening.
* Stricturing type disease with symptoms or signs of non-inflammatory mechanical obstruction or bowel perforation in last 3 months.
* Short bowel syndrome.
* Functional colostomy or ileostomy (note: patients who have had a temporary stoma in the past, which has been reversed, are eligible to enter the study).
* Positive stool laboratory results for enteric pathogens.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 604
Dates: Start 2003-12; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
In the population with CRP ≥ 10 mg/L at baseline
Clinical response at week 6
Clinical response at week 6 and week 26

SECONDARY OUTCOMES:
In the population with CRP ≥ 10 mg/L at baseline - % patients in clinical remission at Week 6; % patients in clinical remission at both Week 6 and Week 26; % patients with IBDQ response at Week 6; % patients with IBDQ response at both Week 6 and Week 2

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma

REFERENCES:
- [Result] Sandborn WJ, Feagan BG, Stoinov S, Honiball PJ, Rutgeerts P, Mason D, Bloomfield R, Schreiber S; PRECISE 1 Study Investigators. Certolizumab pegol for the treatment of Crohn's disease. N Engl J Med. 2007 Jul 19;357(3):228-38. doi: 10.1056/NEJMoa067594. PMID 17634458
- [Result] Rutgeerts P, Schreiber S, Feagan B, Keininger DL, O'Neil L, Fedorak RN; CDP870 Crohn's Disease Study Group. Certolizumab pegol, a monthly subcutaneously administered Fc-free anti-TNFalpha, improves health-related quality of life in patients with moderate to severe Crohn's disease. Int J Colorectal Dis. 2008 Mar;23(3):289-96. doi: 10.1007/s00384-007-0395-7. Epub 2007 Dec 11. PMID 18071721
- [Result] Reilly MC, Gerlier L, Brabant Y, Brown M. Validity, reliability, and responsiveness of the work productivity and activity impairment questionnaire in Crohn's disease. Clin Ther. 2008 Feb;30(2):393-404. doi: 10.1016/j.clinthera.2008.02.016. PMID 18343277
- [Derived] Lewis JD. Anti-TNF antibodies for Crohn's disease--in pursuit of the perfect clinical trial. N Engl J Med. 2007 Jul 19;357(3):296-8. doi: 10.1056/NEJMe078111. No abstract available. PMID 17634466